CLINICAL TRIAL: NCT05194410
Title: The MedMotion Trial on Community Building Through Virtual, Team-Based Exercise and Affects on Physician and Trainee Burnout: A Randomized, Controlled, Multi-Center Trial
Brief Title: The Effect of Community Building Through Virtual, Team-Based Exercise on Burnout
Acronym: MedMotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kerri Palamara McGrath, M.D., Principal Investigator, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000825
Record Dates: First submitted 2021-12-30; First posted 2022-01-18 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Burnout, Professional; Burnout, Student; Community Building; Mentorship; Exercise
Keywords: Burnout, Professional; Burnout, Student; Community Building; Mentorship; Exercise
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 6 months of virtual, team-based exercise
  Interventions: Behavioral: First 3 months of virtual, team-based exercise; Behavioral: Second 3 months of virtual, team-based exercise
- Control (Other): 3 months of usual exercise and then 3 months of virtual, team-based exercise
  Interventions: Behavioral: Second 3 months of virtual, team-based exercise

INTERVENTIONS:
Behavioral: First 3 months of virtual, team-based exercise — Participants will be randomized onto mixed teams of medical students, residents, fellows, and attendings and registered for the virtual, team-based exercise intervention on FitRankings.com. All exercise (including walking, biking, lifting, yoga, and 40+ exercises) will be tracked via user's smartwatches (ie Apple, Garmin), smartphone fitness apps (ie MapMyRun), or manual upload, converted into Metabolic Equivalent of a Task (MET) minutes, and displayed on online leaderboards. Group activities will be encouraged by awarding raffle tickets for prizes to those who submit pictures with their teammates.
  Arms: Intervention
Behavioral: Second 3 months of virtual, team-based exercise — Same as above

SUMMARY:
This study is a randomized controlled trial that will look at whether virtual, team-based exercise improves burnout, sense of community, and mentorship connections among medical students, residents, fellows, and physicians.

DETAILED DESCRIPTION:
Participants will be randomized to either a control group or an intervention group. The intervention group will be further randomized onto teams that will exercise for 3 months. All exercise (including walking, biking, lifting, yoga, and 40+ exercises) will be tracked via user's smartwatches (ie Apple, Garmin), smartphone fitness apps (ie MapMyRun), or manual upload, converted into Metabolic Equivalent of a Task (MET) minutes, and displayed on online leaderboards. Group activities will be encouraged by awarding raffle tickets for prizes to those who submit pictures with their teammates. Primary outcomes will be burnout, sense of community, and mentorship connections, with the hypothesis that getting everyone together for this team-based exercise will improve these metrics. After 3 months, both the control and intervention group will be enrolled in 3 months of the intervention to assess secondary outcomes: long-term burnout, sense of community, and mentorship connections, as well as adherence.

ELIGIBILITY:
Inclusion Criteria:

* Harvard Medical Students (HMS)
* Massachusetts General Hospital (MGH) Residents, Fellows, or Attendings

Exclusion Criteria:

* Non HMS Students or MGH Residents, Fellows, or Attendings

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2021-07-18 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Burnout at 3 months | 0 and 3 months
  Measured via the 2-item Maslach Burnout Inventory (MBI)
  The MBI is a 22-item survey that covers 3 areas: Emotional Exhaustion (EE), Depersonalization (DP), and low sense of Personal Accomplishment (PA). Each subscale includes multiple questions with frequency rating choices of Never, A few times a year or less, Once a month or less, A few times a month, Once a week, A few times a week, or Every day.
  The use of 2 single items from the MBI may also be used. Item 8 ("I feel burned out from my work",) and item 10 ("I have become more callous toward people since I took this job") correlate strongly with the emotional exhaustion and depersonalization subscale scores and concurrent validity has been demonstrated (J Gen Intern Med 2012;27:1445-52. J Gen Inter Med 2009;24:1318-21.)
  Individuals meet burnout criteria if they have high scores on either the EE (total score of 27 or higher) or DP (total score of 10 or higher) subscales.
Change from Baseline Burnout at 6 months | 0 and 6 months
  Measured via the 2-item Maslach Burnout Inventory (MBI)
  The MBI is a 22-item survey that covers 3 areas: Emotional Exhaustion (EE), Depersonalization (DP), and low sense of Personal Accomplishment (PA). Each subscale includes multiple questions with frequency rating choices of Never, A few times a year or less, Once a month or less, A few times a month, Once a week, A few times a week, or Every day.
  The use of 2 single items from the MBI may also be used. Item 8 ("I feel burned out from my work",) and item 10 ("I have become more callous toward people since I took this job") correlate strongly with the emotional exhaustion and depersonalization subscale scores and concurrent validity has been demonstrated (J Gen Intern Med 2012;27:1445-52. J Gen Inter Med 2009;24:1318-21.)
  Individuals meet burnout criteria if they have high scores on either the EE (total score of 27 or higher) or DP (total score of 10 or higher) subscales.
Change in Burnout from 3 to 6 months | 3 and 6 months
  Measured via the 2-item Maslach Burnout Inventory (MBI)
  The MBI is a 22-item survey that covers 3 areas: Emotional Exhaustion (EE), Depersonalization (DP), and low sense of Personal Accomplishment (PA). Each subscale includes multiple questions with frequency rating choices of Never, A few times a year or less, Once a month or less, A few times a month, Once a week, A few times a week, or Every day.
  The use of 2 single items from the MBI may also be used. Item 8 ("I feel burned out from my work",) and item 10 ("I have become more callous toward people since I took this job") correlate strongly with the emotional exhaustion and depersonalization subscale scores and concurrent validity has been demonstrated (J Gen Intern Med 2012;27:1445-52. J Gen Inter Med 2009;24:1318-21.)
  Individuals meet burnout criteria if they have high scores on either the EE (total score of 27 or higher) or DP (total score of 10 or higher) subscales.
Change from Baseline Sense of Community at 3 months | 0 and 3 months
  Measured via the Stanford Professional Fulfillment Index
  The Stanford Professional Fulfillment Index (PFI) is a 16-item survey that covers burnout (work exhaustion and interpersonal disengagement) and professional fulfillment. Response options are on a five-point Likert scale ("not at all true" to "completely true" for professional fulfillment items and "not at all" to "extremely" for work exhaustion and interpersonal disengagement items.)
  Items are scored 0 to 4. Each dimension is treated as a continuous variable. Scale scores are calculated by averaging the item scores of all the items within the corresponding scale. Scale scores can then be multiplied by 25 to create a scale range from 0 to 100. Higher score on the professional fulfillment scale is more favorable while higher scores on the work exhaustion or interpersonal disengagement scales are less favorable.
Change from Baseline Sense of Community at 6 months | 0 and 6 months
  Measured via the Stanford Professional Fulfillment Index
  The Stanford Professional Fulfillment Index (PFI) is a 16-item survey that covers burnout (work exhaustion and interpersonal disengagement) and professional fulfillment. Response options are on a five-point Likert scale ("not at all true" to "completely true" for professional fulfillment items and "not at all" to "extremely" for work exhaustion and interpersonal disengagement items.)
  Items are scored 0 to 4. Each dimension is treated as a continuous variable. Scale scores are calculated by averaging the item scores of all the items within the corresponding scale. Scale scores can then be multiplied by 25 to create a scale range from 0 to 100. Higher score on the professional fulfillment scale is more favorable while higher scores on the work exhaustion or interpersonal disengagement scales are less favorable.
Change in Sense of Community from 3 to 6 months | 3 and 6 months
  Measured via the Stanford Professional Fulfillment Index
  The Stanford Professional Fulfillment Index (PFI) is a 16-item survey that covers burnout (work exhaustion and interpersonal disengagement) and professional fulfillment. Response options are on a five-point Likert scale ("not at all true" to "completely true" for professional fulfillment items and "not at all" to "extremely" for work exhaustion and interpersonal disengagement items.)
  Items are scored 0 to 4. Each dimension is treated as a continuous variable. Scale scores are calculated by averaging the item scores of all the items within the corresponding scale. Scale scores can then be multiplied by 25 to create a scale range from 0 to 100. Higher score on the professional fulfillment scale is more favorable while higher scores on the work exhaustion or interpersonal disengagement scales are less favorable.
Change from Baseline Mentorship Connections at 3 months | 0 and 3 months
  Measured via unvalidated survey
  "How many meaningful relationships would you say you have with [medical students, residents/fellows, attendings]?
  A meaningful relationship could include any of the following: a) someone you'd get coffee/meal with, b) someone you'd be comfortable talking about career/life advice, c) someone you would be comfortable catching up with, etc."
Change from Baseline Mentorship Connections at 6 months | 0 and 6 months
  Measured via unvalidated survey
  "How many meaningful relationships would you say you have with [medical students, residents/fellows, attendings]?
  A meaningful relationship could include any of the following: a) someone you'd get coffee/meal with, b) someone you'd be comfortable talking about career/life advice, c) someone you would be comfortable catching up with, etc."
Change in Mentorship Connections from 3 to 6 months | 3 and 6 months
  Measured via unvalidated survey
  "How many meaningful relationships would you say you have with [medical students, residents/fellows, attendings]?
  A meaningful relationship could include any of the following: a) someone you'd get coffee/meal with, b) someone you'd be comfortable talking about career/life advice, c) someone you would be comfortable catching up with, etc."
Change from Baseline Burnout (Mayo) at 3 months | 0 and 3 months
  Measured via the Mayo Wellbeing Index
  The Mayo Wellbeing Index aims to identify distress in a variety of dimensions (burnout, fatigue, low mental/physical quality of life, depression, anxiety/stress). It has separate medical student, resident/fellow, and physicians versions and is a 7-item instrument with yes/no response categories.
  A total score is calculated by adding the number of 'yes' responses. In a sample of physicians, medical students, and US workers, every one point increase in score resulted in a step-wise increased probability of distress and risk for adverse personal and professional consequence. Score range is 0 to 7, and threshold score to identify individuals in distress is 4 or higher for medical students, 5 or higher for residents, 4 or higher for practicing physicians, and 2 or higher for other US workers.
Change from Baseline Burnout (Mayo) at 6 months | 0 and 6 months
  Measured via the Mayo Wellbeing Index
  The Mayo Wellbeing Index aims to identify distress in a variety of dimensions (burnout, fatigue, low mental/physical quality of life, depression, anxiety/stress). It has separate medical student, resident/fellow, and physicians versions and is a 7-item instrument with yes/no response categories.
  A total score is calculated by adding the number of 'yes' responses. In a sample of physicians, medical students, and US workers, every one point increase in score resulted in a step-wise increased probability of distress and risk for adverse personal and professional consequence. Score range is 0 to 7, and threshold score to identify individuals in distress is 4 or higher for medical students, 5 or higher for residents, 4 or higher for practicing physicians, and 2 or higher for other US workers.
Change in Burnout (Mayo) from 3 to 6 months | 3 and 6 months
  Measured via the Mayo Wellbeing Index
  The Mayo Wellbeing Index aims to identify distress in a variety of dimensions (burnout, fatigue, low mental/physical quality of life, depression, anxiety/stress). It has separate medical student, resident/fellow, and physicians versions and is a 7-item instrument with yes/no response categories.
  A total score is calculated by adding the number of 'yes' responses. In a sample of physicians, medical students, and US workers, every one point increase in score resulted in a step-wise increased probability of distress and risk for adverse personal and professional consequence. Score range is 0 to 7, and threshold score to identify individuals in distress is 4 or higher for medical students, 5 or higher for residents, 4 or higher for practicing physicians, and 2 or higher for other US workers.

SECONDARY OUTCOMES:
Engagement in First Half of Study | 3 months
  Registration of >0 Metabolic Equivalent of a Task (MET) minutes on FitRankings platform
Engagement in Second Half of Study | 6 months
  Registration of >0 Metabolic Equivalent of a Task (MET) minutes on FitRankings platform
Change in Baseline Exercise at 3 months | 0 and 3 months
  On average, how many days per week do you exercise for 30 minutes or more? (0-7 days)
Change in Baseline Exercise at 6 months | 0 and 6 months
  On average, how many days per week do you exercise for 30 minutes or more? (0-7 days)
Change in Exercise from 3 to 6 months | 3 and 6 months
  On average, how many days per week do you exercise for 30 minutes or more? (0-7 days)
Change in Baseline Comfortability at work at 3 months | 0 and 3 months
  How comfortable do you feel about working with [medical students, residents/fellows, attending physicians] at your affiliated hospital?
  (1=not at all, 2=slightly, 3=moderately, 4=very, 5=extremely)
Change in Baseline Comfortability at work at 6 months | 0 and 6 months
  How comfortable do you feel about working with [medical students, residents/fellows, attending physicians] at your affiliated hospital?
  (1=not at all, 2=slightly, 3=moderately, 4=very, 5=extremely)
Change in Comfortability at work from 3 to 6 months | 3 and 6 months
  How comfortable do you feel about working with [medical students, residents/fellows, attending physicians] at your affiliated hospital?
  (1=not at all, 2=slightly, 3=moderately, 4=very, 5=extremely)

CONTACTS AND LOCATIONS:
Overall Officials: Logan Briggs, BA, Study Director — Harvard Medical School (HMS and HSDM)
Locations (2):
- United States (2):
  - Harvard Medical School, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Medicine in Motion Trial Website — https://www.medmotion.org/trial